CLINICAL TRIAL: NCT02658968
Title: A Phase 1 Dose Finding Study of Lutetium (177Lu)-Lilotomab Satetraxetan (Betalutin®) in Patients With Relapsed/Refractory, Diffuse Large B-cell Lymphoma, Not Eligible for Autologous Stem Cell Transplant
Brief Title: Study of Betalutin for Treatment of Relapsed or Refractory Non-Hodgkin Lymphoma (LYMRIT-37-05)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nordic Nanovector (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2015-001933-26
Record Dates: First submitted 2015-12-22; First posted 2016-01-20 (Estimated); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Relapsed, Diffuse Large B-cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
Keywords: Radioimmunotherapy; Lu-177; Phase I study; Betalutin; ARC; Antibody Radionuclide Conjugate; HH1; Rituximab; 177Lu-DOTA-HH1; Lilotomab; Lutetium (177Lu)-lilotomab satetraxetan; Additional relevant MeSH terms:; Lymphoma; Lymphoma, Non-Hodgkin; Immune System Diseases; Immunoproliferative Disorders; Diffuse Large B-Cell Lymphoma; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type; DLBCL; Refractory DLBCL; Relapsed DLBCL
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse; AIDS-Related Complex; Lymphoma; Lymphoma, Non-Hodgkin; Immune System Diseases; Immunoproliferative Disorders; Lymphatic Diseases; Lymphoproliferative Disorders; Neoplasms; Neoplasms by Histologic Type | interventions — tetulomab tetraxetan lu-177; Lutetium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Betalutin (Experimental): 10 MBq/kg b.w., in escalated doses with lilotomab pre-dosing
  Interventions: Drug: Betalutin

INTERVENTIONS:
Drug: Betalutin — Dose finding study, starting on 10 MBq/kg b.w. Betalutin® (lutetium (177Lu)-lilotomab satetraxetan), single injection with lilotomab pre-dosing.
  Other Names: Betalutin, lutetium (177Lu)-lilotomab satetraxetan

SUMMARY:
This study is a phase 1, dose finding, open-label study in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL). This is a dose escalating study to define the maximum tolerated dose (MTD) of lutetium (177Lu)-lilotomab satetraxetan (Betalutin®) in DLBCL patients who are not eligible for autologous stem cell transplant. The study will also assess safety and tolerability, pharmacokinetics, biodistribution and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years.
2. Histologically confirmed DLBCL (WHO classification).
3. Received at least one prior line of therapy including immuno-chemotherapy.
4. In first or subsequent relapse, or refractory to the last treatment (defined as less than a complete metabolic response to the last treatment, or disease progression within 6 months from the last treatment).
5. Not suitable for, or declined/unwilling to undergo intensive therapy, including high dose chemotherapy and autologous stem cell transplantation (ASCT).
6. Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (at least one objectively bi-dimensionally measurable (nodal) lesion (>1.5 cm in its largest dimension by CT scan).
7. Negative human anti-mouse antibody (HAMA) test.
8. Life expectancy of at least 3 months.
9. Bone marrow tumour infiltration <25% tumour cells.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
11. Normal organ and bone marrow function defined as:

    1. Absolute neutrophil count ≥1.5 x 109/L
    2. Platelet count ≥150 x 109/L;
    3. Haemoglobin ≥9 g/dL
    4. Total bilirubin ≤1.5 x upper limit of normal (ULN) (except patients with documented Gilbert's syndrome)
    5. Liver enzymes: Aspartate transaminase (AST); Alanine transaminase (ALT) or Alkaline phosphatase (ALP) ≤2.5 x ULN (or ≤5.0 x ULN if liver involvement by primary disease)
    6. Adequate renal function as demonstrated by a serum creatinine ≤1.5 mg/dL or a creatinine clearance >60 mL/min
    7. Normal coagulation parameters (elevated international normalized ratio (INR), prothrombin time or activated partial thromboplastin time (APTT) ≤1.3 ULN range acceptable)
12. Women of childbearing potential must:

    1. Understand that the study medication may have teratogenic risk
    2. Have a negative serum pregnancy test at screening and before Betalutin injection
    3. Commit to continued abstinence from heterosexual intercourse (excluding periodic abstinence or the withdrawal method) or begin two acceptable methods of birth control with a Pearl-Index ≤ 1%. without interruption from 4 weeks before starting study drug, throughout study drug therapy and for 12 months after end of study drug therapy, even if she has amenorrhoea. Apart from abstinence, acceptable methods of birth control are:

       * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
       * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
       * Intrauterine device (IUD)
       * Intrauterine hormone-releasing system (IUS)
       * Bilateral tubal occlusion
       * Vasectomised partner
13. Male patients must agree to use condoms during intercourse throughout study drug therapy and the following 12 months.
14. Ability to give written, informed consent prior to any study-specific screening procedures, with the understanding that the consent may be withdrawn by the patient at any time without prejudice.
15. Capable of understanding the protocol requirements, is willing and able to comply with the study protocol procedures, and has signed the informed consent document.
16. A negative Hepatitis B test (HBsAg and anti-HBc) and negative HIV test during screening

Exclusion Criteria:

1. Prior hematopoietic allogenic stem cell transplantation.
2. Prior autologous stem cell transplantation.
3. Previous total body irradiation.
4. Prior anti-lymphoma therapy (chemotherapy, immunotherapy or other investigational agent), excluding corticosteroids within 4 weeks prior to start of study treatment (i.e. rituximab) (G-CSF or GM-CSF are permitted up to 2 weeks prior to start of study treatment.)
5. Patients who are receiving any other investigational agents.
6. Patients with known or suspected central nervous system involvement of lymphoma.
7. History of a previous treated cancer except for the following:

   1. Adequately treated local basal cell or squamous cell carcinoma of the skin
   2. Cervical carcinoma in situ
   3. Superficial bladder cancer
   4. Localized prostate cancer undergoing surveillance or surgery
   5. Localised breast cancer treated with surgery and radiotherapy but not including systemic chemotherapy
   6. Other adequately treated Stage 1 or 2 cancer currently in complete remission
8. Pregnant or breastfeeding women.
9. Exposure to another CD37 targeting drug.
10. Allergy to X ray contrast agents.
11. A known hypersensitivity to rituximab, HH1, Betalutin or murine proteins or any excipient used in rituximab, lilotomab or Betalutin.
12. Has received a live attenuated vaccine within 30 days prior to enrolling in the study.
13. Evidence of severe or uncontrolled systemic diseases:

    1. Uncontrolled infection including evidence of ongoing systemic bacterial, fungal, or viral infection (excluding viral upper respiratory tract infections) at the time of initiation of study treatment
    2. Pulmonary conditions e.g. unstable or uncompensated respiratory disease
    3. Hepatic, renal neurological or metabolic conditions - which in the opinion of the investigator would compromise the protocol objectives
    4. Psychiatric conditions e.g. patients unlikely to comply with the protocol, e.g. mental condition rendering the patient unable to understand the nature, scope, and possible consequences of participating in the study
    5. History of erythema multiforme, toxic epidermal necrolysis or Stevens-Johnson syndrome
    6. Cardiac conditions, including:

       * history of acute coronary syndromes (including unstable angina)
       * class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system;
       * known uncontrolled arrhythmias (except sinus arrhythmia) in the past 24 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Illidge, PhD MB BS, Principal Investigator — University of Manchester, The Christie NHS Foundation Trust
Locations (10):
- United States (3):
  - University of California, San Diego (UCSD) - Moores Cancer Center, San Diego, California
  - University of California, San Francisco (UCSF) - Innovation, Technology & Alliances, San Francisco, California
  - Sylvester Comprehensive Cancer Centre, Miami, Florida
- Klinikum rechts der Isar der TU München, Munich, Germany
- Italy (3):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Hospital Universitari i Politècnic La Fe, Valencia, Spain
- United Kingdom (2):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology and Oncology Centre, Bristol
  - Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahle J, Repetto-Llamazares AH, Mollatt CS, Melhus KB, Bruland OS, Kolstad A, Larsen RH. Evaluating antigen targeting and anti-tumor activity of a new anti-CD37 radioimmunoconjugate against non-Hodgkin's lymphoma. Anticancer Res. 2013 Jan;33(1):85-95. PMID 23267131
- [Background] Repetto-Llamazares AH, Larsen RH, Mollatt C, Lassmann M, Dahle J. Biodistribution and dosimetry of (177)Lu-tetulomab, a new radioimmunoconjugate for treatment of non-Hodgkin lymphoma. Curr Radiopharm. 2013 Mar;6(1):20-7. doi: 10.2174/1874471011306010004. PMID 23256748

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened in the 28 days before receiving rituximab (42 days before receiving lilotomab and Betalutin). Participants were then allocated to one of four treatment cohorts following a "3+3" design. They received rituximab on Day -14, followed by Betalutin and lilotomab on Day 0. Two participants received rituximab but were withdrawn prior to receiving lilotomab and Betalutin and were therefore replaced.
Groups:
- 60/10: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 10 MBq/kg, single injection with lilotomab 60 mg/m2 pre-dosing on Day 0 following rituximab pre-treatment on Day -14.
- 100/10: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 10 MBq/kg, single injection with lilotomab 100 mg/m2 pre-dosing on Day 0 following rituximab pre-treatment on Day -14.
- 100/15: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 15 MBq/kg, single injection with lilotomab 100 mg/m2 pre-dosing on Day 0 following rituximab pre-treatment on Day -14.
- 100/20: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 20 MBq/kg, single injection with lilotomab 100 mg/m2 pre-dosing on Day 0 following rituximab pre-treatment on Day -14.
- Rituximab Only: Received rituximab pre-treatment on Day -14. Did not receive Betalutin or lilotomab
Period: Received Rituximab
Arm/Group | 60/10 | 100/10 | 100/15 | 100/20 | Rituximab Only
Started | 3 | 3 | 3 | 7 | 2
Completed | 3 | 3 | 3 | 7 | 0
Not Completed | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 1
Period: Received Lilotomab and Betalutin
Arm/Group | 60/10 | 100/10 | 100/15 | 100/20 | Rituximab Only
Started | 3 | 3 | 3 | 7 | 0
Completed | 0 | 0 | 0 | 1 | 0
Not Completed | 3 | 3 | 3 | 6 | 0
Not completed — Disease progression (including death due to disease progression) | 2 | 0 | 3 | 3 | 0
Not completed — Progressive disease | 1 | 0 | 0 | 0 | 0
Not completed — Start of further anticancer therapy | 0 | 2 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants who received rituximab
Groups:
- Total: Total of all reporting groups
Arm/Group | 60/10 | 100/10 | 100/15 | 100/20 | Rituximab Only | Total
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 2 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (16.09) | 56.7 (10.21) | 77.3 (76.0) | 81.0 (7.07) | 72 (7.07) | 73.5 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 3 | 1 | 9
  Male | 1 | 2 | 1 | 4 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 5 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 5 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 2
ECOG score [Count of Participants; unit: Participants] — 0-5 scale (5 the worst outcome) 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  5. Dead
  Participants
    Score 0 | 0 | 2 | 0 | 3 | 0 | 5
    Score 1 | 2 | 0 | 2 | 3 | 1 | 8
    Score 2 | 1 | 1 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With DLTs to Determine the MTD
Description: To determine the MTD of Betalutin that can be administered to DBLCL patients with lilotomab. The MTD was the highest dose at which less than two out of six participants experienced a dose limiting toxicity (DLT) defined as:
  * Haematologic toxicity:
    * Grade 4 neutropenia observed for greater than 7 days' duration
    * Grade 4 thrombocytopenia observed for greater than 7 days' duration
    * Grade 3 or 4 neutropenia associated with fever (≥38.5°C) of any duration
    * Grade 3 or 4 thrombocytopenia with bleeding
    * Thrombocytopenia with any requirement for more than one platelet transfusion before recovering to Grade 1 or less
    * Grade 4 anaemia, unexplained by underlying disease
  * Non-haematologic toxicity:
    * Grade 3 nausea/vomiting/diarrhoea lasting longer than 72 hours despite maximal care or Grade 4
    * Any other Grade 3 or 4 non-haematologic toxicities
    * Any Grade 3 or 4 electrolyte abnormalities that do not resolve to Grade 1 or baseline within 24 hours
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- 60/10: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 10 MBq/kg, single injection with lilotomab 60 mg/m2 pre-dosing.
- 100/10: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 10 MBq/kg, single injection with lilotomab 100 mg/m2 pre-dosing.
- 100/15: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 15 MBq/kg, single injection with lilotomab 100 mg/m2 pre-dosing.
- 100/20: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 20 MBq/kg, single injection with lilotomab 100 mg/m2 pre-dosing.
Arm/Group | 60/10 | 100/10 | 100/15 | 100/20
Number analyzed (Participants) | 3 | 3 | 3 | 7
Participants | 0 | 0 | 0 | 1

2. Secondary Outcome: The Best Overall Tumour Response
Description: Efficacy evaluations are measured by tumour response rates using CT and PET/CT imaging with responses classified as described in "Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification" (Cheson, 2014). The Cheson criteria, 2014 are a combined score taking into consideration, positive or negative scored PET scan, the contrast enhanced CT images and bone marrow biopsies when available.
Time Frame: 3 months - 2 years
Population: Participants who had a baseline and at least one post-baseline computed tomography scan
Measure: Count of Participants; unit: Participants
Arm/Group | 60/10 | 100/10 | 100/15 | 100/20
Number analyzed (Participants) | 1 | 2 | 2 | 3
Participants
  Progressive disease | 1 | 1 | 1 | 1
  No response/stable disease | 0 | 1 | 0 | 1
  Complete response | 0 | 0 | 1 | 1

3. Secondary Outcome: Dosimetry
Description: Dosimetry will be evaluated by the estimated absorbed radiation dose to target organs.
Time Frame: 3 weeks
Population: Participants having dosimetry evaluation and having the schedule of whole body imaging or SPECT/CT scans
Measure: Number; unit: Gray
Arm/Group | 60/10 | 100/10
Number analyzed (Participants) | 1 | 1
Gray
  Liver | 1.33 | 0.46
  Spleen | 1.39 | 2.63
  Kidneys | 0.70 | 0.73
  Image-based Red Marrow | 0.52 | 0.38
  Total Body | 0.07 | 1.16

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the time of rituximab infusion up to 12 weeks after Betalutin administration on Day 0. Treatment-related adverse events were collected up to 2 years
Description: Treatment emergent adverse events were summarized separately after rituximab and after Betalutin/lilotomab
Groups:
- 60/10: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 10 MBq/kg, single injection with lilotomab 60 mg/m2 .
- 100/10: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 10 MBq/kg, single injection with lilotomab 100 mg/m2.
- 100/15: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 15 MBq/kg, single injection with lilotomab 100 mg/m2 .
- 100/20: Betalutin® (lutetium (177Lu)-lilotomab satetraxetan) 20 MBq/kg, single injection with lilotomab 100 mg/m2 pre-dosing on Day 0.
- Rituximab: Rituximab pre-treatment on Day -14
Arm/Group | 60/10 | 100/10 | 100/15 | 100/20 | Rituximab
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 4/7 | 2/18
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 2/3 | 3/7 | 4/18
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 5/7 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 60/10 (N=3) | 100/10 (N=3) | 100/15 (N=3) | 100/20 (N=7) | Rituximab (N=18)
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 60/10 (N=3) | 100/10 (N=3) | 100/15 (N=3) | 100/20 (N=7) | Rituximab (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 2
Extravasation (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 1 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0
Gamma glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Thoracic outlet syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Vascular compression (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Dysphonea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/68/NCT02658968/Prot_SAP_000.pdf